CLINICAL TRIAL: NCT04707066
Title: Comprehensive Adaptive Multisite Prevention of University Student Suicide (CAMPUS): A Multisite Trial With Duke as a Site, and Duke as Single IRB of Record
Brief Title: Comprehensive Adaptive Multisite Prevention of University Student Suicide
Acronym: CAMPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00103346; Pro00104815 (Other: Duke University IRB); R01MH116062 (NIH); R01MH116052 (NIH); R01MH116050 (NIH); R01MH116061 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Suicide
Keywords: Dialectical Behavior Therapy (DBT); Collaborative Assessment and Management of Suicide (CAMS); Sequential, multiple assignment, randomized trials (SMART); University Students
MeSH Terms: conditions — Suicide | interventions — Therapeutics; Cell Adhesion Molecules; Clinical Trials, Phase I as Topic; Dialectical Behavior Therapy; Clinical Trials, Phase II as Topic; Maintenance

STUDY DESIGN:
Intervention Model Description: Sequential, multiple assignment, randomized trials (SMART) design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Responder, thus placed into ongoing Maintenance/Monitoring.
  Interventions: Behavioral: Treatment As Usual (TAU); Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) - Phase 2
- 2 (Experimental): Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Insufficient Responder, then assigned to Phase 2 CAMS.
  Interventions: Behavioral: Treatment As Usual (TAU); Behavioral: Dialectical Behavior Therapy (DBT) - Phase 2
- 3 (Experimental): Subject assigned to CAMS for Phase 1. Subject is a Phase 1 CAMS Insufficient Responder, then assigned to Phase 2 DBT.
  Interventions: Behavioral: Treatment As Usual (TAU); Behavioral: Maintenance/Monitoring - Phase 2
- 4 (Experimental): Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Responder, thus placed into ongoing Maintenance/Monitoring.
  Interventions: Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) - Phase 1; Behavioral: Dialectical Behavior Therapy (DBT) - Phase 2
- 5 (Experimental): Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Insufficient Responder, then assigned to Phase 2 CAMS.
  Interventions: Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) - Phase 1; Behavioral: Maintenance/Monitoring - Phase 2
- 6 (Experimental): Subject assigned to TAU for Phase 1. Subject is a Phase 1 TAU Insufficient Responder, then assigned to Phase 2 DBT.
  Interventions: Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) - Phase 1; Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) - Phase 2

INTERVENTIONS:
Behavioral: Treatment As Usual (TAU) — Treatment As Usual
  Other Names: TAU - Phase 1
  Arms: 1; 2; 3
Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) - Phase 1 — Collaborative Assessment and Management of Suicidality
  Other Names: CAMS
  Arms: 4; 5; 6
Behavioral: Dialectical Behavior Therapy (DBT) - Phase 2 — Dialectical Behavior Therapy
  Arms: 2; 4
Behavioral: Maintenance/Monitoring - Phase 2 — Maintenance/Monitoring
  Arms: 3; 5
Behavioral: Collaborative Assessment and Management of Suicidality (CAMS) - Phase 2 — Collaborative Assessment and Management of Suicidality (CAMS) - Phase 2
  Arms: 1; 6

SUMMARY:
Suicide is the 2nd leading cause of death among college students and suicidal ideation and suicide-related behaviors are a frequent presenting problem at college counseling centers (CCCs), which are overburdened. Studies show that some students respond rapidly to treatment, whereas others require considerably more resources. Evidence-based adaptive treatment strategies (ATSs) are needed to address this heterogeneity in responsivity and complexity. ATSs individualize treatment via decision rules specifying how the type and intensity of an intervention can be sequenced based on risk factors, response, or compliance.

The purpose of this multisite study is to investigate the effectiveness of four adaptive treatment strategies (ATSs) to treat college students who report suicidal ideation when first seeking services at their college counseling center

This multisite study will enroll moderately to severely suicidal college students in the "emerging adulthood" phase (ages 18-25) seeking services at CCCs. This Sequential Multi-Assignment Randomized Trial (SMART) will have two stages of intervention. In Stage 1, 700 participants from four CCCs will be randomized to 4-8 weeks of: 1) a suicide-focused treatment - Collaborative Assessment and Management of Suicidality (CAMS) or 2) Treatment as Usual (TAU). Sufficient responders to either intervention will discontinue services/be stepped down. Non-responders will be re-randomized to one of two Stage 2 higher intensity/dosage intervention options for an additional 4-16 weeks: 1) CAMS (either continued or administered for the first time) or 2) Comprehensive Dialectical Behavior Therapy (DBT), which includes individual therapy, skills group, and phone/text coaching for the clients and peer consultation for the counselors.

DETAILED DESCRIPTION:
This study will utilize a Sequential Multi-Assignment Randomized Trial (SMART) design. College students seeking counseling services through the College Counseling Centers (CCCs) will be recruited.

In Stage 1, student participants will be initially randomized into either treatment as usual (TAU) or Collaborative Assessment and Management of Suicidality (CAMS). Student participants receiving TAU will receive the customary treatment they would receive at the CCC at a frequency typical to the site (e.g., once a week). Student participants receiving the CAMS intervention will receive CAMS through weekly sessions with a counselor that will last for 50-60 minutes.

Responders to either CAMS or TAU may stop intervention after three consecutive weeks of non-engagement in suicidal acts combined with the ability to cope with suicidal ideation, if present, based on counselor's clinical global impression ratings of improvement and severity. Stage 1 has an intended duration of between 4 and 8 weeks.

Non-responders to Stage 1 treatments, will be re-randomized to one of two Stage 2 treatments: CAMS or Dialectical Behavior Therapy (DBT). Student participants receiving DBT will engage in individual therapy and a skills training group. Stage 2 has an intended treatment duration between 4 and 16 weeks.

All treatment in Stage 1 and Stage 2 (TAU, CAMS, and DBT) will usually be administered in person.

Counselors will provide TAU, CAMS, and DBT to study participants. They will also participate in CAMS and DBT trainings and ongoing consultation teams for each.

The project estimates 36 months (3 years) total duration from beginning of recruitment until final data collection.

The duration of treatment will vary from 4 to 24 weeks and is based on response. Total participant duration in study, due to the assessments, is approximately 48 weeks (which includes the 24-week follow-up assessment).

Counselor participants will participate for 1-3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled at the university;
2. 18 to 25 years of age;
3. Moderate to severe SI over the last two weeks indicated by a score of ³2 on the Counseling Center Assessment of Psychological Symptoms (CCAPS-34) question, "I have thoughts of ending my life" (range is 0 "not at all like me" to 4 "extremely like me"); and
4. Agree to video recording of all therapy and assessment sessions.

Exclusion Criteria:

1. Students who are deemed clinically inappropriate to receive services at the CCC by an intake counselor because of imminent risk, severe psychosis, or inability to remain enrolled in school (e.g., academic failure);
2. Students being unable to remain on campus long enough to go through the minimum number of sessions for Stage 1 (4 sessions);
3. Students who have received services at the CCC within the last three months (i.e., ATSs must be based on a new treatment episode).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 227 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Suicide Ideation - Stage 1 | Baseline to the end of Stage 1 treatment (up to 8 weeks)
  Change in score of CAMS Scale for Suicidal Ideation (SSI). This is a 19 question measure, each rated from 0-2. Total score is from 0-38, with a higher score indicating greater suicidality concern.
Suicide Ideation - Stage 2 | Baseline to the end of Stage 2 treatment (up to 20 weeks)
  Change in score of CAMS Scale for Suicidal Ideation (SSI). This is a 19 question measure, each rated from 0-2. Total score is from 0-38, with a higher score indicating greater suicidality concern.
Suicide Ideation - 6 month follow-up | Baseline to 6 month follow-up
  Change in score of CAMS Scale for Suicidal Ideation (SSI). This is a 19 question measure, each rated from 0-2. Total score is from 0-38, with a higher score indicating greater suicidality concern.
Non-Suicidal Self Injury - Stage 1 | To the end of Stage 1 treatment (up to 8 weeks)
  Total Occurrences of Non-Suicidal Self Injury
Non-Suicidal Self Injury - Stage 2 | To the end of Stage 2 treatment (up to 20 weeks)
  Total Occurrences of Non-Suicidal Self Injury
Non-Suicidal Self Injury - 6 month follow-up | To 6 month follow-up
  Total Occurrences of Non-Suicidal Self Injury
Suicide Attempts - Stage 1 | To the end of Stage 1 treatment (up to 8 weeks)
  Total Occurrences of Suicide Attempts
Suicide Attempts - Stage 2 | To the end of Stage 2 treatment (up to 20 weeks)
  Total Occurrences of Suicide Attempts
Suicide Attempts - 6 month follow-up | To 6 month follow-up
  Total Occurrences of Suicide Attempts

CONTACTS AND LOCATIONS:
Overall Officials: Scott Compton, PhD, Principal Investigator — Duke University; Jacqueline Pistorello, PhD, Principal Investigator — University of Nevada at Reno (UNR); Shireen Rizvi, PhD, Principal Investigator — Rutgers University; John Seeley, PhD, Principal Investigator — University of Oregon
Locations (4):
- United States (4):
  - University of Nevada - Reno, Reno, Nevada
  - Rutgers University, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina
  - University of Oregon, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: Yes
We will participant de-identified data (linked only by GUID) with the National Institute of Mental Health Data Archive (NDA). The NDA is an informatics system and research data repository developed by the National Institutes of Health (NIH) to share research data. The NDA provides the infrastructure to store, search across, and analyze various types of data. In addition, The NDA provides longitudinal storage of a research participant's information generated by one or more research studies. In other words, the NDA is able to associate a single research participant's genomic, imaging, clinical assessment and other information even if the data were collected at different locations or through different studies. By doing so, the NDA gives researchers access to more data than they can collect on their own, making it easier and faster for researchers to gather, evaluate, and share research information from a variety of sources.
Supporting Information: Study Protocol, SAP
Time Frame: All subject data will be submitted for inclusion in the NDA, through the conclusion of data collection activities. Data is to be submitted cumulatively, every 6 months.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Qualified researchers who have completed a Data Use Certification and received approval from the NDA Data Access Committee (DAC) may be approved to access broadly shared data. A separate request process exists for access to data in federated sources. Additionally, the DAC and support staff at NIH have access to NDA shared data.
URL: https://nda.nih.gov/nda/about-us.html

REFERENCES:
- [Derived] Blalock K, Pistorello J, Rizvi SL, Seeley JR, Kassing F, Sinclair J, Oshin LA, Gallop RJ, Fry CM, Snyderman T, Jobes DA, Crumlish J, Krall HR, Stadelman S, Gozenman-Sapin F, Davies K, Steele D, Goldston DB, Compton SN. The Comprehensive Adaptive Multisite Prevention of University Student Suicide Trial: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 22;14:e68441. doi: 10.2196/68441. PMID 40262131

DOCUMENTS (1):
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04707066/ICF_000.pdf